CLINICAL TRIAL: NCT06156813
Title: Validity and Reliability of Turkish Version of the Lower Extremity Motor Activity Log
Brief Title: Turkish Lower-Extremity Motor Activity Log (LE-MAL)
Status: Recruiting | Type: Observational
Sponsor: Gaziantep Islam Science and Technology University (Other)
Responsible Party: Sponsor
Other Study IDs: ipek.kirmaci
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Stroke; Spastic Paraplegia
Keywords: LE-MAL; Spasticity; Measurement; validity; reliability
MeSH Terms: conditions — Stroke; Paraplegia; Muscle Spasticity | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Diagnostic test — Measurements for validity and reliability

SUMMARY:
The Motor Activity Log was developed to measure paretic upper extremity use in daily activities in the real-life context (real world) of people with different health conditions, including stroke. Subsequently, the Lower Extremity Motor Activity Diary was developed. This survey is a semi-structured survey in which the participant is asked to rate himself/herself according to each scale over 14 activities.

DETAILED DESCRIPTION:
The Motor Activity Log was developed to measure paretic upper extremity use in daily activities in the real-life context (real world) of people with different health conditions, including stroke. Real-world use outside the individual's clinical/laboratory environment, including daily activities (e.g., walking indoors and outdoors above ground, climbing stairs, getting in and out of a car, jumping over an object, picking up an object, sitting and standing) It's about what they do.

The Motor Activity Log is a reliable patient self-report measure and correlates significantly with another real-world measure, the accelerometer.

Adaptation of the Motor Activity Log to the lower extremity involved the development of three subscales to measure changes in types of activity that are bilateral in nature and use of the paretic lower extremity: level of assistance, functional ability, and confidence. The Lower Extremity Motor Activity Log is a semi-structured questionnaire in which the participant is asked to rate himself on each scale across 14 activities. The score for each scale is the average of the rate provided for each activity. Additionally, a composite score can be calculated that combines all scales through assistance, functional ability, and confidence scores.

A preliminary study with individuals with stroke using the English version of the Lower Extremity Motor Activity Log-14 showed that the total score was 0.93, 0.90, 0.94, and 0.88 test-retest for the composite score, assistance, functional ability, and confidence scales, respectively. The test showed that it has reliability.

The aim of this study is to investigate the reliability and validity of the Turkish version of the Lower Extremity Motor Activity Log-14.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 18-80 living in Gaziantep who applied to the neurology outpatient clinic of Hospital and were diagnosed with stroke.

Exclusion Criteria:

* Patients with a history of trauma within the last year, alcohol and substance addiction, and pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Tr- LE-MAL | baseline and two weeks later
  t is a semi-structured interview that includes questions to determine the participant's level of assistance, movement quality and confidence while performing a 14-day activity.

SECONDARY OUTCOMES:
Stroke Impact Scale | Baseline
  This scale, which aims to evaluate the perception of the quality of life after stroke by the patients themselves or their caregivers, consists of 8 subsections and 59 questions.
6 min walk test | Baseline
  Functional capacity in terms of mobility is evaluated by measuring the person's maximum walking distance within a six-minute period.

CONTACTS AND LOCATIONS:
Overall Officials: Zekiye İpek Katırcı Kırmacı, Principal Investigator — Gaziantep Islam Science and Technology University
Locations (1):
- Gaziantep Islam Science and Technology University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided